CLINICAL TRIAL: NCT05336643
Title: Pelvic Side Wall Lymph Node Detection in Rectal Cancer Using Dual Radioisotope and Fluorescence Guidance
Brief Title: Radioisotope and Fluorescence Guidance in Rectal Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 147974; 307317 (Other: IRAS)
Record Dates: First submitted 2022-03-30; First posted 2022-04-20 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Rectal Cancer; Lymph Node Metastasis
MeSH Terms: conditions — Rectal Neoplasms; Lymphatic Metastasis

STUDY DESIGN:
Intervention Model Description: Open label, single arm, feasibility study for a medical device
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radioisotope and fluorescence guidance (Experimental): Patients undergoing curative resection for rectal cancer will receive a peritumoural, submucosal administration of indocyanine green and technetium-99m nanocolloid. Intraoperatively the SENSEI gamma probe and Da Vinci Firefly will be used to identify pelvic side wall lymph nodes.
  Interventions: Device: Radiofluorescence

INTERVENTIONS:
Device: Radiofluorescence — Assessment of pelvic sidewall with Firefly and Sensei

SUMMARY:
A study to investigate if pelvic side wall lymph nodes that remain after neo-adjuvant chemoradiotherapy can be identified intraoperatively using dual radioisotope and fluorescence guidance.

DETAILED DESCRIPTION:
Background Total mesorectal excision (TME) revolutionised the management of rectal cancer by improving outcomes and standardising surgical technique. When excising mesorectal lymph nodes, most involved nodes are removed. However, a proportion of lower rectal lymphatic drainage is through the pelvic sidewall (PSW) system, all PSW nodes are left behind in TME. Up to 15% patients with rectal cancer have PSW involvement at presentation, this is associated with increased local recurrence.

Problem There are two main approaches in the management of PSW nodes. In the Western hemisphere, patients are typically staged with pre-operative MRI. Those with nodes undergo neo-adjuvant chemoradiotherapy to downstage the tumour, followed by surgical resection, PSW lymph nodes are left in place. In the East patients undergo PSW lymph node dissection at the time of rectal resection. There is evidence that lymphadenectomy at initial surgery or after chemoradiotherapy improves oncological outcome, though this is at the cost of increased morbidity, worsening urinary and sexual function.

Objective The aim is to make PSW lymph node dissection safer and more targeted. This initial feasibility study, is investigating if PSW lymph nodes can be individually identified using dual modalities, fluorescence, and a radioisotope tracer. The fluorophore indocyanine green (ICG) has been used successfully for lymph node mapping in rectal cancer. ICG and Technetium-99m nanocolloid (Tc99m), a radioisotope, have been used as dual tracers for lymph nodes in gynaecological, esophagogastric and oral surgery, but never in rectal surgery.

Method The investigators have designed an open label, single-centre, feasibility study to investigate if PSW lymph nodes can be identified intra-operatively using a radioisotope and fluorescence. Ten post neo-adjuvant chemotherapy rectal cancer patients will be scheduled for resection. Pre-operatively patients will receive an injection of Tc99m and ICG to the submucosa around the tumour. Patients will undergo single-photon emission computed tomography (SPECT) scanning to identify lymphatic drainage. Intra-operatively, after bowel resection, the surgical team will examine the PSW for lymph nodes using a minimally invasive gamma probe (SENSEI, Lightpoint Medical) to detect Tc99m, and a near infrared camera system (Firefly, Intuitive) to visualise ICG. The primary outcome is intraoperative detection of PSW lymph nodes.

Significance The aim from this feasibility study is to demonstrate that individual PSW nodes can be detected intra-operatively. By proving this technique, the investigators will design a larger study to investigate the oncological outcome of excising individual involved nodes, with the aim of reducing PSW recurrence and surgical morbidity.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Primary diagnosis of biopsy-proven rectal cancer
* Scheduled for curative robotic surgery of primary tumour
* Have signed an approved informed consent form for the study
* Be willing and able to comply with the study protocol

Exclusion Criteria:

* Known allergy or history of adverse reaction to Technetium-99m nanocolloid or indocyanine green
* Pregnant or lactating subjects
* Subjects who, in the Investigator's and/or designee's opinion, have any medical condition that makes the subject a poor candidate for the investigational procedure, or interferes with the interpretation of study results

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Lymph node detection with indocyanine green and near-infrared light source | 12 months
  Intraoperative identification of pelvic side wall lymph nodes using fluorescence. After resection of the rectal specimen the near infrared light source will be switched on and the pelvic side wall will be assessed for lymph nodes seen on SPECTCT. Primary outcome will be recorded as "yes" or "no".
Lymph node detection with technetium 99m colloid and SENSEI gamma probe | 12 months
  Intraoperative identification of pelvic side wall lymph nodes using radioisotope. After resection of the rectal specimen the gamma probe will be switched on and the pelvic side wall will be assessed for lymph nodes seen on SPECTCT. Primary outcome will be recorded as "yes" or "no".

SECONDARY OUTCOMES:
Radioactive count of identified lymph nodes (MBq) | 12 months
  Usability of drop in gamma probe - effectiveness 1
  Intraoperative identification of pelvic side wall lymph nodes using radioisotope. After resection of the rectal specimen the gamma probe will be switched on and the pelvic side wall will be assessed for lymph nodes seen on SPECTCT.
  Secondary outcome is the gamma radiation count of identified nodes recorded in megabecquerel (MBq)
Background radioactive count (MBq) | 12 months
  Usability of drop in gamma probe - effectiveness 2
  Intraoperative identification of pelvic side wall lymph nodes using radioisotope. After resection of the rectal specimen the gamma probe will be switched on and the pelvic side wall will be assessed for lymph nodes seen on SPECTCT.
  Secondary outcome is the gamma radiation count of background radiation, measured underneath camera port, pointing up towards port, recorded in megabecquerel (MBq)
Time to lymph node identification (seconds) | 12 months
  Usability of drop in gamma probe - effectiveness 3
  Intraoperative identification of pelvic side wall lymph nodes using radioisotope. After resection of the rectal specimen the gamma probe will be switched on and the pelvic side wall will be assessed for lymph nodes seen on SPECTCT.
  Secondary outcome is time taken for lymph node identification, recorded in seconds
Usability of drop in probe (System usability scale) | 12 months
  Usability of drop in gamma probe - satisfaction
  Intraoperative identification of pelvic side wall lymph nodes using radioisotope. After resection of the rectal specimen the gamma probe will be switched on and the pelvic side wall will be assessed for lymph nodes seen on SPECTCT.
  Secondary outcome is the usability of the SENSEI gamma probe using the System Usability Scale (Score 0-100)
Lymph nodes identified on SPECTCT | 12 months
  In the morning patients receive a peritumoral submucosal injection of technetium 99m nano colloid. After a 4 hour interval they undergo SPECTCT.
  Number of lymph nodes identified on SPECTCT.
Concordance of nodes seen on PET MRI/CT and SPECTCT | 12 months
  In the lead up to surgery (>24 hours prior) patients will undergo PET MRI/CT. In the morning patients receive a peritumoral submucosal injection of technetium 99m nano colloid. After a 4 hour interval they undergo SPECTCT.
  Percentage of nodes seen on PET MRI/CT seen on SPECTCT (%)

CONTACTS AND LOCATIONS:
Overall Officials: Simon Wan, Principal Investigator — University College London Hospitals
Locations (1):
- University College London Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
As this is a small pilot study there is no plan to publish IPD. However, if requested by researchers then it can be shared.
Supporting Information: CSR
Time Frame: Data will be available after completion of the study. In line with University protocols data is stored for 20 years.
Access Criteria: Other researchers for systematic review and meta-analysis